CLINICAL TRIAL: NCT00002129
Title: A Phase I Study of Three Doses of OPC-8212 (Vesnarinone) in HIV-Infected Persons With CD4+ Cell Number > 300 Cells/mm3
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka America Pharmaceutical (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 234A; 22-93-251
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1996-04

CONDITIONS: HIV Infections
Keywords: vesnarinone
MeSH Terms: conditions — HIV Infections | interventions — vesnarinone

INTERVENTIONS:
Drug: Vesnarinone

SUMMARY:
To examine the safety and tolerance of three doses of oral vesnarinone in HIV-infected patients with CD4 count > 300 cells/mm3.

DETAILED DESCRIPTION:
Twelve patients per dose level receive vesnarinone at 1 of 3 doses for 12 weeks. At least six patients at a given dose level must have completed 2 weeks of treatment before dose is escalated in subsequent patients.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Chemoprophylaxis for Pneumocystis carinii, candida, mycobacteria, and herpes simplex.

Patients must have:

* Asymptomatic HIV infection.
* CD4 count > 300 cells/mm3.
* No prior AIDS-defining illness or current constitutional symptoms of HIV disease.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Current history of cardiac disease, including patients who exhibit long QT syndrome on EKG screening.
* Active malignancy other than cutaneous basal cell carcinoma or in situ carcinoma of the cervix.

Concurrent Medication:

Excluded:

* Antiretroviral agents, including ddI, ddC, and AZT.
* Immunosuppressive agents.
* Investigational HIV drugs/therapies including vaccines.
* Interferon.
* Steroids (other than topical).
* Hematopoietins.
* Megestrol acetate.
* Trimethoprim/sulfamethoxazole in excess of 160 mg trimethoprim and 800 mg sulfamethoxazole thrice weekly.
* Cytotoxic chemotherapy.

Concurrent Treatment:

Excluded:

* Radiation therapy.

Patients with the following prior conditions are excluded:

* Prior history of cardiac disease.
* History of agranulocytosis or severe (grade 3) drug-induced neutropenia or documented abnormalities in granulocyte number or function.

Prior Medication:

Excluded:

* AZT, ddI, and ddC within 14 days prior to study entry.
* Prior cytotoxic chemotherapy.

Prior Treatment:

Excluded:

* Radiation therapy (including electron beam irradiation) within 30 days prior to study entry.

Active illicit drug abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA School of Medicine, Los Angeles, California, United States

REFERENCES:
- [Background] Mitsuyasu R, Bort L, Miles SA, Hardy WD, Petit RG. Preliminary results of a phase I study of vesnarinone (OPC-8212) in HIV-infected persons with CD4 > 300 cells/MM3. Int Conf AIDS. 1994 Aug 7-12;10(1):8 (abstract no 005B)